CLINICAL TRIAL: NCT00322465
Title: Phase II Randomized, Placebo-Controlled Double-Blind 4-Arm Trial for the Treatment of Non-Gonococcal Urethritis (NGU): Doxycycline (Plus or Minus Tinidazole) Versus Azithromycin (Plus or Minus Tinidazole)
Brief Title: NGU: Doxycycline (Plus or Minus Tinidazole) Versus Azithromycin (Plus or Minus Tinidazole)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-0120
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2011-05

CONDITIONS: Urethritis
Keywords: non-gonococcal urethritis, doxycycline, azithromycin, sexually transmitted, tinidazole
MeSH Terms: conditions — Urethritis | interventions — Tinidazole; Doxycycline; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Doxycycline (Experimental): Doxycycline 100 mg orally twice daily (2 pills/day = 200 mg/day) for 7 days plus placebo azithromycin orally single dose and placebo tinidazole.
  Interventions: Other: Placebo; Drug: Doxycycline
- Doxycycline + Tinidazole (Experimental): Doxycycline 100 mg orally twice daily for 7 days plus placebo azithromycin single dose plus tinidazole 2 gm orally single dose (4 tablets at 500 mg each).
  Interventions: Drug: Tinidazole; Other: Placebo; Drug: Doxycycline
- Azithromycin (Experimental): Azithromycin 1 gram (gm) orally single dose (2 tablets at 500 milligrams (mg) each) plus doxycycline placebo twice daily for 7 days plus tinidazole placebo single dose.
  Interventions: Other: Placebo; Drug: Azithromycin
- Azithromycin + Tinidazole (Experimental): Azithromycin 1 gm orally single dose (2 tablets at 500 mg each) plus doxycycline placebo twice daily for 7 days plus tinidazole single dose (4 tablets at 500 mg each).
  Interventions: Drug: Tinidazole; Other: Placebo; Drug: Azithromycin

INTERVENTIONS:
Drug: Tinidazole — 2 gm single dose (4 tablets orally at 500 mg each).
  Arms: Azithromycin + Tinidazole; Doxycycline + Tinidazole
Other: Placebo — Placebo capsule will be filled with lactose only and be identical in appearance to the capsule of Azithromycin, Tinidazole, Doxycycline.
Drug: Doxycycline — 100 mg orally, twice daily for 7 days.
  Arms: Doxycycline; Doxycycline + Tinidazole
Drug: Azithromycin — 1 gram (gm) (2 tablets orally at 500 milligrams (mg) each).
  Arms: Azithromycin; Azithromycin + Tinidazole

SUMMARY:
This study will look at the safety, effectiveness, and tolerability of combination medications for the initial treatment of non-gonococcal urethritis (NGU). NGU is inflammation of the tube that carries urine from the bladder. NGU is caused by bacteria that may be passed from person to person during sex. This study will compare the 2 currently recommended NGU treatments, doxycycline and azithromycin, taken with tinidazole (another medication to treat certain sexually transmitted infections). Tinidazole used with doxycycline or azithromycin may cure NGU better than when doxycycline or azithromycin is used alone. Study participants will be 300 men ages 16-45 years with NGU attending sexually transmitted disease clinics in Birmingham, AL; New Orleans, LA; Durham, NC; and Baltimore, MD. Study participation will last 7 weeks and involve 3 visits. At each visit, participants will provide a urine sample, have 2 urethral swabs, and have their urethra checked for discharge indicating infection.

DETAILED DESCRIPTION:
This study represents a clinical evaluation of the use of combination therapy for the initial treatment of non-gonococcal urethritis (NGU). This study will provide more current data on the comparison of cure rates between the 2 currently recommended therapies for NGU, doxycycline and azithromycin. Emerging clinical data has suggested that the latter may have become more efficacious for NGU as it is more effective in eradicating Mycoplasma (M.) genitalium from the genital tract than the former. Only in vitro data, limited as it is, suggests that doxycycline should be active against M. genitalium. The researchers hypothesize that cure rates for NGU will be significantly improved for both doxycycline and azithromycin using combination therapy with tinidazole. Important safety and tolerability data will be collected with regards to the use of combination therapy. Additionally, the study will provide data on the prevalence of the targeted pathogens in 4 geographic areas and on characteristics of men with NGU that may help to target populations who would benefit the most from combination therapy. The researchers hypothesize that currently recommended initial therapies for NGU are inadequate in at least certain populations due to lack of coverage for Trichomonas (T.) vaginalis. The researchers further hypothesize that between the 2 currently recommended regimens, azithromycin will result in a greater number of cures than doxycycline due to its greater efficacy in M. genitalium infected men. The primary study objectives are to: compare the clinical cure rates of doxycycline versus doxycycline with tinidazole; and azithromycin versus azithromycin with tinidazole for the treatment of NGU; and to evaluate the safety and tolerability of doxycycline/tinidazole and azithromycin/tinidazole in the treatment of NGU. Secondary study objectives are to: evaluate microbiological cure of Chlamydia (C.) trachomatis, T. vaginalis, M. genitalium in men treated with doxycycline versus doxycycline with tinidazole; and azithromycin versus azithromycin with tinidazole. Analysis will also include: (doxycycline plus doxycycline/tinidazole) versus (azithromycin plus azithromycin/tinidazole); for the clinical cure rates, analysis will also include: (doxycycline plus doxycycline/tinidazole) versus (azithromycin plus azithromycin/tinidazole); determine the prevalence of C. trachomatis, T. vaginalis, and M. genitalium in the study population of men with non-gonococcal urethritis; determine clinical, behavioral, and demographic predictors of the above organisms in men with non-gonococcal urethritis; and collect specimens for future studies to determine the role of unique and novel pathogens in the etiology of non-gonococcal urethritis. Outcome measures include clinical failure, clinical cure, microbiological cure, and unevaluable cure assessed at the first and second follow-up visits. Study participants will include 300 men ages 16-45 years with NGU attending sexually transmitted disease clinics in Birmingham, AL; New Orleans, LA; Durham, NC; and Baltimore, MD. Subjects will be randomly assigned to 1 of 4 active treatment arms: 75 subjects doxycycline; 75 subjects doxycycline plus tinidazole; 75 subjects azithromycin; and 75 subjects azithromycin plus tinidazole.

ELIGIBILITY:
Inclusion Criteria:

* Male, 16 to 45 years old.
* Symptoms of non-gonococcal urethritis (NGU), including urethral discharge and/or dysuria for less than or equal to 14 days, or urethral discharge on exam.
* Urethral smear with greater than or equal to 5 polymorphonuclear leukocytes (PMNs) per 3-5 oil immersion fields.
* Willing to abstain from sexual intercourse or use condoms during the study.
* Willingness to provide written consent.

Exclusion Criteria:

* Presence of gonorrhea at baseline visit.
* History of recurrent non-gonococcal urethritis (NGU) (3 or more episodes in the prior year) or history of recent NGU (within past 30 days).
* Signs or symptoms of epididymitis or prostatitis.
* Known allergy to or intolerance of tinidazole, tetracyclines, macrolides or metronidazole.
* History of photosensitivity related to doxycycline use.
* Received systemic antibiotics within 30 days of study enrollment.
* Unwillingness to abstain from alcohol for 24 hours after enrollment.
* Serious underlying infection, including known HIV or other primary or secondary immunosuppression.
* Concomitant infection, which requires antimicrobial therapy.
* History of mental illness, which would preclude responsible participation in the study.
* Current drug abuse that might affect ability to follow the protocol.
* Previously enrolled in this study.
* Men who have sex with men, due to different microbiology of NGU.
* Voided within the previous hour.
* Ingested alcohol within the past 8 hours.
* Subject requires concurrent lithium, anticoagulation therapy, or antabuse.

Ages: 16 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 305 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - Delgado Personal Health Center, New Orleans, Louisiana
  - Johns Hopkins Hospital - Emergency Medicine, Baltimore, Maryland
  - University of North Carolina School of Medicine - Center for Infectious Diseases, Chapel Hill, North Carolina

REFERENCES:
- [Result] Schwebke JR, Rompalo A, Taylor S, Sena AC, Martin DH, Lopez LM, Lensing S, Lee JY. Re-evaluating the treatment of nongonococcal urethritis: emphasizing emerging pathogens--a randomized clinical trial. Clin Infect Dis. 2011 Jan 15;52(2):163-70. doi: 10.1093/cid/ciq074. PMID 21288838

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline: Doxycycline 100 mg by mouth twice a day (2 pills/day = 200 mg/day) for 7 days plus placebo azithromycin by mouth single dose and placebo tinidazole.
- Doxycycline + Tinidazole: Doxycycline 100 mg by mouth twice a day for 7 days plus placebo azithromycin single dose plus tinidazole 2 gm by mouth single dose (4 tablets at 500 mg each).
- Azithromycin: Azithromycin 1 gm by mouth single dose (2 tablets at 500 mg each) plus doxycycline placebo twice a day for 7 days plus tinidazole placebo single dose.
- Azithromycin + Tinidazole: Azithromycin 1 gm by mouth single dose (2 tablets at 500 mg each) plus doxycycline placebo twice a day for 7 days plus tinidazole single dose (4 tablets at 500 mg each).
Period: Overall Study
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Started | 76 (Randomized) | 73 (Randomized) | 77 (Randomized) | 79 (Randomized)
Completed | 56 (Second follow-up visit or clinical failure at first follow-up visit) | 49 (Second follow-up visit or clinical failure at first follow-up visit) | 51 (Second follow-up visit or clinical failure at first follow-up visit) | 53 (Second follow-up visit or clinical failure at first follow-up visit)
Not Completed | 20 | 24 | 26 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole | Total
Number analyzed (Participants) | 76 | 73 | 77 | 79 | 305
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2 | 3 | 7
  Between 18 and 65 years | 75 | 72 | 75 | 76 | 298
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7.0) | 27.8 (6.8) | 26.4 (6.7) | 25.7 (7.2) | 26.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 76 | 73 | 77 | 79 | 305
Region of Enrollment [Number; unit: participants]
  United States | 76 | 73 | 77 | 79 | 305

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Doxycycline/Tinidazole and Azithromycin/Tinidazole: Number of Participants Reporting Nausea
Description: At all study visits, unsolicited adverse events were recorded. Nausea, Vomiting, Abdominal pain, and Diarrhea were recorded using National Cancer Institute Common Toxicity Criteria (Version 3.0).
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: Modified intent-to-treat population was comprised of all subjects randomized who received at least one dose of study drug therapy or placebo
Measure: Number; unit: Participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Participants | 3 | 4 | 0 | 4

2. Primary Outcome: Safety and Tolerability of Doxycycline/Tinidazole and Azithromycin/Tinidazole: Number of Participants Reporting Vomiting
Description: as for outcome 1
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Participants | 4 | 2 | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving Clinical Cure of NGU With (Doxycycline Plus Doxycycline/Tinidazole) Versus (Azithromycin Plus Azithromycin/Tinidazole)
Description: Clinical Cure of NGU: Did not meet criteria for clinical failure at last evaluable follow-up visit.
  Clinical Failure at first follow-up: [Persistent symptoms AND >= 5 PMNs per 3-5 oil immersion fields (regardless of urethral discharge)] OR Persistent urethral discharge on exam (regardless of symptoms or number of PMNs).
  Clinical Failure at second follow-up: >= 5 PMNs per 3-5 oil immersion fields (regardless of symptoms or presence of urethral discharge) OR Persistent urethral discharge on exam (regardless of symptoms or number of PMNs)
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Doxycycline + (Doxycycline + Tinidazole): Doxycycline 100 mg PO BID (2 pills/day = 200 mg/day) for 7 days plus placebo azithromycin PO single dose and placebo tinidazole + (Doxycycline 100 mg PO BID for 7 days plus placebo azithromycin single dose plus tinidazole 2 gm PO single dose (4 tablets at 500 mg each)).
- Azithromycin + (Azithromycin + Tinidazole): Azithromycin 1 gm PO single dose (2 tablets at 500 mg each) plus doxycycline placebo BID for 7 days plus tinidazole placebo single dose + (Azithromycin 1 gm PO single dose (2 tablets at 500 mg each) plus doxycycline placebo BID for 7 days plus tinidazole single dose (4 tablets at 500 mg each))
Arm/Group | Doxycycline + (Doxycycline + Tinidazole) | Azithromycin + (Azithromycin + Tinidazole)
Number analyzed (Participants) | 149 | 156
Percentage of participants | 49 | 44

4. Secondary Outcome: Percentage of Participants Achieving Microbiological Cure of Chlamydia Trachomatis With Doxycycline Versus Doxycycline With Tinidazole; and Azithromycin Versus Azithromycin With Tinidazole
Description: Microbiological cure of Chlamydia trachomatis refers to the percentage of men with NGU who were negative for Chlamydia trachomatis at the last available result and had been positive for Chlamydia trachomatis at baseline.
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: Participants who were positive at baseline, returned for follow-up, and had evaluable test results.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 34 | 24 | 26 | 25
Percentage of participants | 89 | 75 | 66 | 61

5. Secondary Outcome: Percentage of Participants Achieving Microbiological Cure of Trichomonas Vaginalis With Doxycycline Versus Doxycycline With Tinidazole; and Azithromycin Versus Azithromycin With Tinidazole
Description: Microbiological cure of Trichomonas vaginalis refers to the percentage of men with NGU who were negative for Trichomonas vaginalis (swab and urine specimens) at the last available result and had been positive for Trichomonas vaginalis at baseline (swab or urine specimen).
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: Participants who were positive at baseline, returned for follow-up, and had evaluable test results.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 9 | 9 | 7 | 5
Percentage of participants | 55 | 75 | 56 | 50

6. Secondary Outcome: Percentage of Participants Achieving Microbiological Cure of Mycoplasma Genitalium With Doxycycline Versus Doxycycline With Tinidazole; and Azithromycin Versus Azithromycin With Tinidazole
Description: Microbiological Cure of Mycoplasma Genitalium refers to the percentage of men with NGU who were negative for Mycoplasma Genitalium at the last available result and had been positive for Mycoplasma Genitalium at baseline.
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: Participants who were positive at baseline, returned for follow-up, and had evaluable test results.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 21 | 18 | 22 | 23
Percentage of participants | 23 | 32 | 52 | 68

7. Secondary Outcome: Prevalence of Chlamydia Trachomatis in Men With Non-gonococcal Urethritis
Description: Percentage of men with non-gonococcal urethritis that had a positive result for Chlamydia trachomatis at baseline (enrollment)
Time Frame: Baseline (enrollment visit)
Population: All study participants with evaluable baseline test results.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Percentage of participants | 50 | 38 | 38 | 46

8. Secondary Outcome: Prevalence of Trichomonas Vaginalis (Swab or Urine Specimen) in Men With Non-gonococcal Urethritis
Description: Percentage of men with non-gonococcal urethritis that had a positive result for Trichomonas vaginalis from a urethral swab or urine specimen at baseline (enrollment)
Time Frame: Baseline (enrollment visit)
Population: All study participants with evaluable baseline test results.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Percentage of participants | 14 | 16 | 12 | 10

9. Secondary Outcome: Prevalence of Mycoplasma Genitalium in Men With Non-gonococcal Urethritis
Description: Percentage of men with non-gonococcal urethritis that had a positive result for Mycoplasma genitalium at baseline (enrollment)
Time Frame: Baseline (enrollment)
Population: All study participants with evaluable baseline test results.
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 76 | 79
Percentage of participants | 29 | 30 | 32 | 32

10. Secondary Outcome: Clinical, Behavioral, and Demographic Predictors of Chlamydia Trachomatis in Men With Non-gonococcal Urethritis
Description: Clinical, behavioral, and demographic variables considered were discharge amount and appearance; condom use last sex; new recent partner; number of partners and new partners in last 30 days as well as last 3 months; number of times vaginal sex, oral sex, or anal sex in past 30 days; always/almost always used condom in last 3 months.
Time Frame: Baseline (enrollment visit)
Population: All study participants who met major eligibility criteria (per protocol) with evaluable baseline measures.
Measure: Number; unit: Participants
Arm/Group | All Participants Analyzed
Number analyzed (Participants) | 290
Participants
  Positive for Chlamydia Trachomatis at Baseline | 128
  Negative for Chlamydia Trachomatis at Baseline | 162
Statistical Analysis 1: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for age (per 5 years) is 1 versus the alternative that it is greater than or less than 1. This was tested in a multivariable logistic regression model; Test type: Superiority or Other; p = 0.005, Regression, Logistic — A priori threshold for statistical significance was p<0.05; Odds ratio has been adjusted for other independent variables included in the model, which are found in the other Statistical Analysis sections; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.60 to 0.91]
Statistical Analysis 2: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for scant discharge (reference category is no discharge) is 1 versus the alternative that it is greater than or less than 1. This was tested in a multivariable logistic regression model; Test type: Superiority or Other; p = 0.780, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.33 to 2.30]
Statistical Analysis 3: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for moderate discharge amount (reference category is no discharge) is 1 versus the alternative that it is greater than or less than 1. This was tested in a multivariable logistic regression model; Test type: Superiority or Other; p = 0.164, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.75 to 5.33]
Statistical Analysis 4: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for large amount of discharge (reference category is no discharge) is 1 versus the alternative that it is greater than or less than 1. This was tested in a multvariable logistic regression model; Test type: Superiority or Other; p = 0.919, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.23 to 5.17]
Statistical Analysis 5: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for 2 or more sex partners in the last 3 months (reference category is 0-1 partners) is 1 versus the alternative that it is greater than or less than 1; Test type: Superiority or Other; p = 0.051, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.00 to 3.30]
Statistical Analysis 6: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for 1 or more new sex partners in the last 30 days (reference category is 0) is 1 versus the alternative that it is greater than or less than 1; Test type: Superiority or Other; p = 0.076, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 4.42, 95% CI 2-sided [0.86 to 22.74]
Statistical Analysis 7: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for ever having sex with a prostitute or sex for money, drugs, or other things (reference category is no) is 1 versus the alternative that it is greater than or less than 1; Test type: Superiority or Other; p = 0.075, Regression, Logistic — A priori threshold fors tatistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.13 to 1.10]
Statistical Analysis 8: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for visit due to sexually transmitted disease contact (reference category is no) is 1 versus the alternative that it is greater than or less than 1; Test type: Superiority or Other; p < 0.001, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 3.92, 95% CI 2-sided [1.93 to 7.98]

11. Secondary Outcome: Clinical, Behavioral, and Demographic Predictors of Trichomonas Vaginalis in Men With Non-gonococcal Urethritis
Description: Trichomonas vaginalis was determined from urethral swab or urine specimen. Clinical, behavioral, and demographic predictors considered included discharge amount and appearance; condom use last sex; new recent partner; number of partners and new partners in last 30 days and last 3 months; number of times vaginal sex, oral sex, or anal sex in last 30 days; always/almost always used condom in last 3 months.
Time Frame: Baseline (enrollment visit)
Population: All study participants who met major eligibility criteria (per protocol) with evaluable baseline results.
Measure: Number; unit: Participants
Arm/Group | All Participants Analyzed
Number analyzed (Participants) | 291
Participants
  Positive for Trichomonas Vaginalis at Baseline | 38
  Negative for Trichomonas Vaginalis at Baseline | 253
Statistical Analysis 1: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for 2 or more sex partners in the last 3 months (reference category is 0-1 partners) is 1 versus the alternative that it is greater than or less than 1. This was tested in a multivariable logistic regression model; Test type: Superiority or Other; p = 0.009, Regression, Logistic — A priori threshold for statistical significance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 0.20, 95% CI 2-sided [0.06 to 0.66]
Statistical Analysis 2: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for ever having sex with a prostitute or for money, drugs, or other things(reference category is no) is 1 versus the alternative that it is greater than or less than 1. This was tested in a multivariable logistic regression model; Test type: Superiority or Other; p = 0.074, Regression, Logistic — A priori threshold for statistical signficance was p<0.05; [statistical method as in outcome 10, analysis 1]; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.92 to 6.22]

12. Secondary Outcome: Clinical, Behavioral, and Demographic Predictors of Mycoplasma Genitalium in Men With Non-gonococcal Urethritis
Description: Logistic multiple regression with independent variable selection based on single variable models with p<0.10. Participants positive at enrollment for Mycoplasma genitalium from urine specimen. Potential variables: discharge amount and appearance; condom use last sex; new recent partner, number of partners and new partners in last 30 days and last 3 months; number of times vaginal sex, oral sex, or anal sex in last 30 days; always/almost always used condom last 3 months.
Time Frame: Baseline (enrollment visit)
Population: All study participants who met major eligibility criteria (per protocol) with evaluable baseline results.
Measure: Number; unit: Participants
Arm/Group | All Participants Analyzed
Number analyzed (Participants) | 292
Participants
  Positive for Mycoplasma Genitalium at Baseline | 90
  Negative for Mycoplasma Genitalium at Baseline | 202
Statistical Analysis 1: Comparison: All Participants Analyzed; The null hypothesis is that the odds ratio for age (per 5 years) is 1 versus the alternative that the odds ratio is greater than or less than 1; Test type: Superiority or Other; p = 0.032, Regression, Logistic — A priori threshold for statistical significance was p<0.05; No other independent variables were included in the model; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.66 to 0.98]

13. Primary Outcome: Safety and Tolerability of Doxycycline/Tinidazole and Azithromycin/Tinidazole: Number of Participants Reporting Stomach Upset
Description: At all study visits, unsolicited adverse events were recorded.
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Participants | 1 | 1 | 1 | 0

14. Primary Outcome: Safety and Tolerability of Doxycycline/Tinidazole and Azithromycin/Tinidazole: Number of Participants Reporting of Abdominal Pain
Description: as for outcome 1
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Participants | 6 | 5 | 3 | 5

15. Primary Outcome: Safety and Tolerability of Doxycycline/Tinidazole and Azithromycin/Tinidazole: Number of Participants Reporting Diarrhea
Description: as for outcome 1
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Participants | 0 | 3 | 3 | 7

16. Primary Outcome: Percentage of Participants Achieving Clinical Cure of Non-gonococcal Urethritis (NGU) With Doxycycline Versus Doxycycline With Tinidazole; and Azithromycin Versus Azithromycin With Tinidazole
Description: Clinical Cure of NGU: Did not meet criteria for clinical failure at last evaluable follow-up visit.
  Clinical Failure at first follow-up: [Persistent symptoms AND >= 5 polymorphonuclear leukocytes (PMNs) per 3-5 oil immersion fields (regardless of urethral discharge)] OR Persistent urethral discharge on exam (regardless of symptoms or number of PMNs).
  Clinical Failure at second follow-up: >= 5 PMNs per 3-5 oil immersion fields (regardless of symptoms or presence of urethral discharge) OR Persistent urethral discharge on exam (regardless of symptoms or number of PMNs)
Time Frame: First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Population: Modified intent to treat: all subjects randomized who received at least one dose of study drug therapy or placebo
Measure: Number; unit: Percentage of participants
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Number analyzed (Participants) | 76 | 73 | 77 | 79
Percentage of participants | 47 [40.8 to 64.2] | 51 [37.4 to 61.3] | 39 [49.3 to 72.0] | 48 [40.4 to 63.3]

17. Secondary Outcome: Specimens for Future Studies to Determine the Role of Unique and Novel Pathogens in the Etiology of Non-gonococcal Urethritis
Description: Urethral swabs and urine specimens collected at each study visit for future studies to determine the role of unique and novel pathogens in the etiology of non-gonococcal urethritis
Time Frame: Baseline (enrollment); First follow-up visit (Day 15-19), second follow-up visit (Day 35-45)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Trial involved an enrollment visit, first follow-up visit (Day 15-19), and second follow-up visit (Day 35-45). Timeframe was approximately 7 weeks.
Description: Adverse events were unsolicited.
Arm/Group | Doxycycline | Doxycycline + Tinidazole | Azithromycin | Azithromycin + Tinidazole
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/73 | 0/77 | 0/79
Other Adverse Events (participants affected / at risk) | 18/76 | 25/73 | 11/77 | 24/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=76) | Doxycycline + Tinidazole (N=73) | Azithromycin (N=77) | Azithromycin + Tinidazole (N=79)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (5) | 3 (3) | 5 (5)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloody discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital Herpes (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital lesion (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Genital pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 0 (0) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Light headedness/ dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (7) | 4 (4) | 0 (0) | 4 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory infection/ respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus infection/ sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spider bite/ anthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stomach upset/ stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste abnormality/ disgeusia (Nervous system disorders) | 0 (0) | 6 (6) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Wrist sprain/ joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No